CLINICAL TRIAL: NCT01201070
Title: Effects of the Administration Of Antithrombin on the Coagulation Status and on the Inflammatory Response in Patients With Low Plasmatic Levels of Antithrombin After Cardiac Surgery
Brief Title: Study of Administration Of Antithrombin in Patients With Low Plasmatic Levels of Antithrombin After Cardiac Surgery
Acronym: ATIII
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bari (Other)
Responsible Party: Department of Emergency and Organ Transplant, Division of Cardiac Surgery, University of Bari, Italy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Antithrombin III
Record Dates: First submitted 2010-09-08; First posted 2010-09-14 (Estimated); Last update posted 2010-09-15 (Estimated); Status verified 2010-07

CONDITIONS: Aortic Valve Insufficiency; Aortic Valve Stenosis; Mitral Valve Insufficiency; Mitral Valve Stenosis; Acute Coronary Syndrome
MeSH Terms: conditions — Aortic Valve Insufficiency; Aortic Valve Stenosis; Mitral Valve Insufficiency; Mitral Valve Stenosis; Acute Coronary Syndrome | interventions — Antithrombin III

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- control group (No Intervention)
- no treatment (No Intervention)
- TREATMENT WITH ANTITHROMBIN (Active Comparator): 3000 IU bolus at the time of randomization vs the study group 1000 IU after 8 h (24 h G0) 1000 IU after 16 h (8 h G1) TOTAL 5000/UI 24h
  Interventions: Drug: antithrombin III

INTERVENTIONS:
Drug: antithrombin III — 3000 IU bolus at the time of randomization vs the study group 1000 IU after 8 h (24 h G0) 1000 IU after 16 h (8 h G1) TOTAL 5000/UI 24h
  Arms: TREATMENT WITH ANTITHROMBIN

SUMMARY:
General and specific objectives of the search: evaluate the effects of the administration of Antithrombin III (ATIII) on the activation of the coagulation system and of the fibrinolysis, platelet function, inflammatory response and markers of organ damage in patients undergoing cardiac surgery by cardiopulmonary bypass (CPB) with low plasma levels of post-operative Antithrombin (AT).

ELIGIBILITY:
Inclusion Criteria:

* All patients were candidates for cardiac surgery intervention in extracorporeal circulation

Exclusion Criteria:

* positive history for allergic reactions to AT III
* cardiac surgery "Off-Pump"
* administration of AT during surgery or within 48 h
* treatment with drugs and non-steroidal steroids within 48 h prior
* disorders of coagulation
* platelets <30,000
* pre-existing IRC in dialysis treatment
* severe liver failure
* enlistment in another trial in the last 30 days
* hypothermia
* emergency
* reopening
* length of CEC> 180 minutes
* subjects incapable of giving legal consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with reduced bleeding, transfusion requirements and need of reintervention for bleeding as a measure of efficacy. | until 5 days after surgey

SECONDARY OUTCOMES:
Number of participants with infection as a measure of safety. | until 5 days after surgery
Number of participants with delirium as a measure of safety. | until 5 days after surgery
Number of participants with wound complication as a measure of safety. | until 5 days after surgery
Number of participants with multi organ failure as a measure of safety. | until 5 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Domenico Paparella, Investigator, Principal Investigator — Department of Emergency and Organ Transplant, Division of Cardiac Surgery. University of Bari, Italy
Locations (1):
- Azienda Ospedaliero-Universitaria Policlinico, Bari, Italy